CLINICAL TRIAL: NCT00799123
Title: Urine NT-proBNP Levels and Echocardiographic Findings in Very Low Birth Weight (VLBW) Infants
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Charite University, Berlin, Germany, Department of Neonatology
Other Study IDs: EA2/072/08/2
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Infant, Premature; Ductus Arteriosus, Patent; Ventricular Function, Left
Keywords: NT-proBNP
MeSH Terms: conditions — Premature Birth; Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to evaluate urine NT-proBNP levels and new Echocardiographic Findings in VLBW infants. The investigators hypothesize that high urine NT-proBNP concentrations are associated with a hemodynamically significant ductus arteriosus. The investigators also hypothesized that new echocardiographic parameters such as isovolumic relaxation time (IVRT)is useful for the prediction of ductus intervention.

DETAILED DESCRIPTION:
Urine samples were collected within 24 to 48 hours of age, on day 7, on day 14 and on day 28 of life. The samples were spun and the platelet-free urine was stored at -80°C until NT-proBNP analysis. The NT-proBNP assay was performed with an automated immunoassay (Roche Diagnostics). Color Doppler and tissue Doppler echocardiography was determined at the same time as the urine collection. New echo parameters such as IVRT, tissue velocity, strain and strain rate were measured and compared with the standard parameters for significant ductus arteriosus. Furthermore we compared the tissue Doppler measurements with clinical findings.

ELIGIBILITY:
Inclusion Criteria:

* Written parental informed consent
* VLBW infants
* Admitted to our NICU within 48 hours after birth

Exclusion Criteria:

* No written parental informed consent
* Congenital heart disease
* Death

Ages: 24 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: VLBW infants
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Czernik, MD, Principal Investigator — Charite, Medical University Berlin
Locations (1):
- Charite, Medical University, Berlin, State of Berlin, Germany